CLINICAL TRIAL: NCT00003713
Title: A Phase I, Pharmacokinetic, and Treatment Duration and Escalation Study of Intravenous Intoplicine Administered as a 5 to 21-Day Continuous Infusion Every 4 Weeks
Brief Title: Chemotherapy in Treating Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Purpose: Treatment
Other Study IDs: CDR0000066821; ILEX-INTO101-A6; ILEX-INTO101-A5; SACI-IDD-97-02; UTHSC-9785011033; NCI-V98-1507
Record Dates: First submitted 1999-11-01; First posted 2004-05-03 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2001-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — intoplicine

INTERVENTIONS:
Drug: intoplicine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of intoplicine in treating patients who have advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the intolerable dose level of intoplicine in patients with locally advanced or metastatic cancer. II. Determine recommended phase II dose of intoplicine in these patients. III. Determine the principal and dose limiting toxicities of intoplicine in these patients, and determine the duration and reversibility of the toxicities. IV. Determine the magnitude of plasma concentrations that are achieved and maintained on this regimen and relate this parameter to toxicity outcome and antitumor activity. V. Determine preliminary evidence of antitumor activity of intoplicine in these patients.

OUTLINE: This is a dose escalation study. The first 3 patients receive intoplicine IV by continuous infusion for 5 days. Treatment is repeated every 28 days in the absence of disease progression or unacceptable toxicity. Subsequent cohorts of 3-6 patients receive escalating doses of intoplicine, first by increasing the number of days that the drug is infused to 10, 15, and 21, then by increasing the dosage and keeping the infusion time constant at 21 days. The intolerable dose level is defined as the lowest dose at which at least 2 of 3 or 6 patients experience dose limiting toxicity during course 1 or 2.

PROJECTED ACCRUAL: A total of 20-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven solid tumor refractory to conventional cytotoxic anticancer therapy or for which no curative therapy exists Measurable or evaluable disease No active, progressive brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT/SGPT no greater than 3 times upper limit of normal No nonmalignant hepatic disease Renal: Creatinine no greater than 2.0 mg/dL Potassium and magnesium at least lower limit of normal (LLN) Calcium at least LLN Cardiovascular: QTc interval on echocardiogram less than 450 milliseconds No myocardial infarction within past 6 months No uncontrolled congestive heart failure No unstable angina No active cardiomyopathy No unstable ventricular arrhythmia No uncontrolled hypertension Other: Not pregnant or nursing Fertile patients must use effective contraception Must have functional central venous access device or percutaneous intravenous catheter No known hypersensitivity to intoplicine or its analogs No active alcoholism or drug addiction No uncontrolled, unstable psychotic disorders No serious infections No underlying medical conditions that may be aggravated by treatment

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) and recovered No other concurrent antineoplastic therapy Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy (except short courses (no greater than 5 fractions) of nonmyelosuppressive, palliative radiotherapy) and recovered No concurrent radiotherapy Surgery: Not specified Other: At least 3 weeks since prior investigational therapy No other concurrent investigational therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 1997-08

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - San Antonio Cancer Institute, San Antonio, Texas
- Princess Margaret Hospital, Toronto, Ontario, Canada